CLINICAL TRIAL: NCT03417414
Title: Does CMV Induced Changes in NK Lymphocyte Biology Influence the Effectiveness of Antibody Therapy Used to Treat B Cell Lymphoproliferative Diseases?
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: GNK Cells in CLL and NHL
Record Dates: First submitted 2017-12-15; First posted 2018-01-31 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: B Cell Lymphocytic Leukemia; B Cell Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Leukemia, B-Cell; Lymphoma, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The CMV status of individuals will be measured by serology in the laboratory of Dr. Lee.
  The presence and function of g-NK cells will be identified and quantified following staining with appropriate fluorescent monoclonal antibody conjugates using flow cytometry of peripheral blood.
  Samples from individuals will be examined to determine changes over time associated with remission-induction and maintenance anti-CD20 based treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- B-CLL: Patients with B-Cell CLL
- B-NHL: Patients with B-Cell NHL

SUMMARY:
This is an observational cohort study of patients with a new diagnosis of B cell Chronic Lymphocytic Leukemia or B cell Non-Hodgkin's Lymphoma who will receive an anti-CD20 monoclonal antibody treatment during the induction phase of their treatment. Throughout the study, patients will have four blood draws at specified time points throughout the study. The initial blood draw will be analysed test patients for Cytomegalovirus and conduct a g-NK cell analysis. The final three blood draws will be conducted to analyse the g-NK cells at specified time points. The objectives of this study are to: 1) characterize the frequency of CMV (+) and g-NK (+) individuals in the B-NHL and B-CLL populations, 2) Determine changes in circulating g-NK cells during and after anti-CD20 monoclonal antibody containing remission induction chemotherapy and 3) Evaluate whether the presence of g-NK cells improve the outcome of anti-CD20 monoclonal antibody containing remission induction treatment of patients with B-NHL or B-CLL.

DETAILED DESCRIPTION:
CMV infection results in a unique population of highly effective ADCC effector cells (g-NK) in more than 50% of individuals. Unlike most NK cells, g-NK cells are long-lived and persist for years following primary infection. The g-NK population enlarges following antibody binding through their Fc receptors (FcR) and target engagement by the antibody. The addition of rituximab and other monoclonal antibodies directed against B lymphocyte targets to remission-induction therapy has improved the depth and durability of response for patients with B cell lymphoproliferative diseases, such as Non-hodgkin's lymphoma (NHL) and chronic lymphocytic leukemia (CLL). The effects of rituximab and other monoclonal anti-cancer antibodies are at least partially mediated through ADCC mechanisms.

The purpose of this study is to examine the clinically relevant aspects of g-NK biology during antibody-containing therapy of lymphoproliferative diseases including whether the presence of g-NK might correlate with improved treatment responses.

Up to 160 patients with either B cell NHL or CLL will be enrolled in this study.

The study enrollment will occur over approximately 2 years. Patients will only be involved in this study until their blood samples are collected at the time point described below.

The following data will be abstracted from the clinical record over the course of the study:

* Age (at beginning of remission-induction therapy)
* Gender
* Weight and height
* Pathological diagnosis including subtype and genetic testing when available.
* Stage at diagnosis
* Prognostic index score (IPI or FLIPI as appropriate)
* Date that remission-induction therapy begins
* Chemotherapy used for remission-induction.
* Dose of anti-CD20 antibody administered during remission-induction
* Remission status after 3 cycles of remission-induction therapy (if available)
* Details of maintenance therapy (drug, dose, schedule)
* Date of progression or relapse.

ELIGIBILITY:
Inclusion Criteria:

* New diagnosis of CD20 expressing B-NHL or CLL

  o Up to 1/3rd of enrolled patients may have CLL. Enrollment of patients with CLL will be halted if this criterion is reached.
* Will receive an anti-CD20 monoclonal antibody treatment (including rituximab, obinatuzumab) during the induction phase of treatment
* Has not previously received cytotoxic chemotherapy medications
* Able to provide informed consent

Exclusion Criteria:

* Comorbidities or frailty that would limit estimated survival to <1 year.
* Will not receive active anti-CD20 containing remission induction therapy.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a new diagnosis of CD20 expressing B-NHL or CLL who will receive an anti-CD20 monoclonal antibody treatment during the induction phase of treatment who have not previously been exposed to cytotoxic chemotherapy medications.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Is the presence of gNK cells associated with better clinical responses in rituxan treated lymphoma patients? | 2 years
  Blood samples will be collected at 4 specified time points from each participant.

SECONDARY OUTCOMES:
Are circulating gNK cells capable of killing CD20+ lymphoma cells through rituximab mediated ADCC mechanisms. | 2 years
  Blood samples will be collected at 4 specified time points from each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Harold Atkins, MD FRCP C, Principal Investigator — The Ottawa Hospital

IPD SHARING:
Plan to Share IPD: No